CLINICAL TRIAL: NCT05251415
Title: Constitution of a Collection of Biological Samples With the Aim of Carrying Out Clinico-biological and Pathophysiological Investigations of Systemic Autoimmune Diseases
Brief Title: Clinico-biological Collection to Investigate the Physiopathology of Systemic Autoimmune Diseases
Acronym: ESSAi
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0505
Record Dates: First submitted 2022-01-24; First posted 2022-02-22 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Lupus Erythematosus; Scleroderma; Myositis; Vasculitis; Inflammatory Bowel Diseases
Keywords: systemic autoimmune diseases; scleroderma; lupus; myositis; vasculitis; Inflammatory Bowel Diseases; new therapies
MeSH Terms: conditions — Scleroderma, Diffuse; Myositis; Vasculitis; Inflammatory Bowel Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients suffering from autoimmune disease: Biological samples will be collected in the normal diagnosis and follow-up process. Only blood will be taken in larger quantity.
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood will be taken in larger quantity.

SUMMARY:
The aim of this project is to start a biological and clinical collection of patients presenting systemic autoimmune disease. This collection will provide appropriate biological samples to identify new biomarkers and to be accessible to the medical, scientific and industrial communities for the identification of new therapeutic strategies

DETAILED DESCRIPTION:
Autoimmune diseases group together less than a hundred different clinical entities which are for the most part rare pathologies but which, in combination, concern 5-8% of the adult population with a strong female predominance (FAI²R: the disease chain rare autoimmune and auto-inflammatory drugs, fai2r.org). The common denominator of all these diseases is based on the breakdown of self-tolerance which is the origin of self-reactivity and whose physiopathological mechanisms are still not fully understood, which generates numerous cross-sectional or fundamental studies. In addition to this complexity, there are significant inter-individual variabilities which lead to the definition of subgroups of patients on the basis of the clinical-biological profile and / or the response to treatments. Consequently and in view of the need to establish the diagnosis early and then to propose the best treatment in the perspective of an individualized medicine, the clinical, biological and genetic characteristics of these subgroups of patients must be explored in order to improve diagnostic and therapeutic capacities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rare systemic autoimmune diseases (lupus, scleroderma, myositis for example),
* Patients with atypical presentations of documented or probable systemic autoimmune diseases,
* Patients receiving, or likely to receive new, innovative therapies (new molecule on the market, gene therapy, cell therapy, etc.).

Exclusion Criteria:

* Known anemia and hemoglobin <10 g / dl
* Patients under protective supervision (guardianship, curators)
* Pregnant or breastfeeding woman

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with autoimmune diseases
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2027-04-04 (Estimated); Study Completion 2032-04-04 (Estimated)

PRIMARY OUTCOMES:
Constitution of a collection of biological samples and clinical-biological data from patients with autoimmune diseases | through study completion, an average of 1 year
  Prospective collection of all available biological samples and clinical data collected during the normal clinical care

SECONDARY OUTCOMES:
Identification and / or validation of new biomarkers for diagnostic and / or prognostic purposes | through study completion, an average of 1 year
  Use of immune cells and / or biological liquids obtained from patients for cohort studies with new methods of screening (microarray, flow cytometry)
Identification and / or validation of new predictive biomarkers of relapse and / or response to treatment | through study completion, an average of 1 year
  Use of immune cells and / or biological liquids obtained from patients for cohort studies with new methods of screening (microarray, flow cytometry)
Identification of specificities in these patients in order to improve the diagnosis, treatment decisions and / or the pathophysiological understanding of these diseases | through study completion, an average of 1 year
  Use of immune cells and / or biological samples for transcriptomic and / or proteomic studies, or in order to be used in experimental animal models
Identification of the determinants of immune reconstitution after cell therapy | through study completion, an average of 1 year
  Exploring blood cell populations before and after cell therapy with flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Chloé BOST, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Purpan University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No